CLINICAL TRIAL: NCT00444327
Title: Observational Study of Cord Blood Single Nucleotide Polymorphisms of Genes Related to Atopy and Allergic Diseases
Brief Title: Use Cord Blood Single Nucleotide Polymorphism to Predict the Later Development of Atopy and Allergy
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Min-Sheng General Hospital (Other)
Collaborators: National Taiwan University Hospital (Other)
Responsible Party: Chien-Han Chen, Min-Sheng General Hospital
Other Study IDs: 2007005
Record Dates: First submitted 2007-03-06; First posted 2007-03-07 (Estimated); Last update posted 2009-05-14 (Estimated); Status verified 2009-05

CONDITIONS: Atopy; Allergic Disease
Keywords: single nucleotide polymorphism

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The aim of our study was firstly to detect in cord bloods the polymorphism of genes related to atopy and allergic diseases and to examine their mutual interaction and their associations with cord blood IgE and cytokines. After that, in the prospective follow-up visits, we liked to investigate if the measurement of cord blood SNPs of genes related to atopy and allergic diseases was helpful in predicting the development of atopy and allergic diseases later in life.

ELIGIBILITY:
Inclusion Criteria:

* Apgar score of 5 minutes not less than 7 gestational age not less than 36 weeks

Exclusion Criteria:

* Apgar score of 5 minutes < 7 gestational age < 36 weeks

Max Age: 1 Minute | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: hospital and primary care clinic based study
Sampling Method: Non-Probability Sample
Enrollment: 900 (Estimated)
Dates: Start 2007-03

CONTACTS AND LOCATIONS:
Overall Officials: Chien-Han Chen, M.D., Principal Investigator — Min-Sheng General Hospital
Locations (1):
- Min-Sheng General Hospital, Taoyuan District, Taiwan